CLINICAL TRIAL: NCT00927238
Title: A Pivotal, Multi-Center, Clinical Trial Evaluating The Safety And Effectiveness of The Lumbar TDR Device In Patients With Single-Level Lumbar Degenerative Disc Disease
Brief Title: XL TDR® eXtreme Lateral Total Disc Replacement for the Treatment of Lumbar Degenerative Disc Disease (DDD)
Acronym: XL TDR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NuVasive (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NUVA-LTDR-0701
Record Dates: First submitted 2009-06-22; First posted 2009-06-24 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Degenerative Disc Disease
Keywords: Single Level; Lumbar Disc Disease; DDD
MeSH Terms: conditions — Intervertebral Disc Degeneration; Intervertebral disc disease | interventions — Total Disc Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- XL TDR (Experimental): The XL TDR is indicated for reconstruction of the disc following discectomy in skeletally mature subjects with symptomatic degenerative disc disease (DDD) of the lumbar spine at one level from L1-L5. DDD is defined as discogenic back pain with degeneration of the disc confirmed by patient history radiographic studies.
  Interventions: Device: XL TDR; Other: Lumbar fusion surgery
- Outcomes from lumbar fusion study (Other)
  Interventions: Other: Lumbar fusion surgery

INTERVENTIONS:
Device: XL TDR — This will be a lateral approach discectomy and reconstruction with the insertion of the XL TDR device.
  Other Names: Total disc replacement
  Arms: XL TDR
Other: Lumbar fusion surgery — Lumbar fusion surgery

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of XL TDR in patients with single-level degenerative disc disease compared to other devices approved by the FDA for the same or similar indications.

DETAILED DESCRIPTION:
The XL TDR® eXtreme Lateral Total Disc Replacement consists of two endplates that are provided in a number of sizes to accommodate a variety of patient anatomies and pathologies. The XL TDR device is made up of a ball and socket articulation and the joint is made of CoCrMo alloy.

The XL TDR is intended to be used to reconstruct the spine following the removal of part or all of the intervertebral disc on one level of the lumbar spine.

The XL TDR is indicated for reconstruction of the disc following discectomy in skeletally mature subjects with symptomatic degenerative disc disease (DDD) of the lumbar spine at one level from L1-L5. DDD is defined as discogenic back pain with degeneration of the disc confirmed by patient history radiographic studies.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years of age (inclusive and skeletally mature) at the time of surgery
* Diagnosis of image-confirmed symptomatic DDD at one of the following levels: L1/L2, L2/L3, L3/L4, or L4/L5
* DDD diagnosed using patient history and image-confirmation such as (but not limited to), MRI, CT, or CT Myelogram with one or more of the following factors: contained herniated nucleus pulposus, facet joint degeneration/changes, decreased disc height >2mm, and/or scarring/thickening of ligamentum flavum, annulus fibrosis, or facet joint capsule
* Preoperative ODI ≥ 30 points
* Unresponsive to conservative treatment for ≥ 6 months

Exclusion Criteria:

* Symptomatic multilevel lumbar degeneration
* Chronic back or leg pain of unknown etiology
* Non-contained or extruded herniated nucleus pulpous
* Previous or other lumbar surgery at any level except prior discectomy, laminotomy, or nucleolysis at the same level
* Involved vertebral endplates dimensionally smaller than 45mm in the medial-lateral and/or 20mm in the anterior/posterior directions
* Idiopathic scoliosis
* Defect in the pars interarticularis
* Radiographic signs of significant instability at operative level
* Lytic spondylolisthesis or degenerative spondylolisthesis > than grade 1
* Bony lumbar spinal stenosis
* Radiographic confirmation of significant facet joint disease or degeneration
* Another lumbar device implanted
* Clinically compromised vertebral bodies at the affected level due to trauma
* Presence of metastases or active spinal tumor malignancy
* Osteopenia, osteoporosis, or metabolic bone disease
* Active local or systemic infection, including AIDS and hepatitis
* Rheumatoid arthritis or other autoimmune disease
* Taking any medications or supplements which potentially interfere with bone/soft tissue healing
* Progressive neuromuscular disease
* Allergy to device materials, specifically: cobalt-chromium-molybdenum alloy, titanium, and hydroxyapatite
* BMI >40
* Pregnant, or may become pregnant within follow-up period of study
* Enrolled in another investigational study within the last 90 days
* Waddell signs of inorganic behavior ≥3
* History of substance abuse
* Involved in active spinal litigation
* Receiving workman's compensation for spinal condition
* Mentally incompetent
* Incarcerated
* Unwilling or unable to comply with all protocol visits/assessments

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2009-07; Primary Completion 2014-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Improvement in ODI | December 2012

SECONDARY OUTCOMES:
Disc Height | December 2012

CONTACTS AND LOCATIONS:
Overall Officials: William D Smith, MD, Principal Investigator — Western Regional Center for Brain and Spine Surgery
Locations (17):
- United States (17):
  - Silicon Valley Spine Institute, Campbell, California
  - Conejo Orthopaedic and Spine Institute, Thousand Oaks, California
  - Spine Colorado / Durango Orthopedic Associates, Durango, Colorado
  - Christiana Spine Center, Newark, Delaware
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - South Florida Spine Institute, Miami Beach, Florida
  - Southeastern Spine Center & Research Institute, Sarasota, Florida
  - University of South Florida, Tampa, Florida
  - West Augusta Spine Specialists, Augusta, Georgia
  - Spine Institute of Louisiana, Shreveport, Louisiana
  - Spine Midwest, Jefferson City, Missouri
  - Western Regional Spine Center for Brain and Spine Surgery, Las Vegas, Nevada
  - Buffalo Spine Surgery, Lockport, New York
  - Southern Oregon Orthopedics, Medford, Oregon
  - Southeastern Spine Institute, Mt. Pleasant, South Carolina
  - Central Texas Spine Institute, Austin, Texas
  - Northwest Orthopaedic Specialists, Spokane, Washington